CLINICAL TRIAL: NCT01871480
Title: An Open-label, Randomized, Controlled Study of Gefitinib Plus Autologous Cytokine-Induced Killer Cell Immunotherapy（CIK）Versus Gefitinib Alone As Second Or Third-Line Treatment in Patients With Advanced Adenocarcinoma Non-Small Cell Lung Cancer
Brief Title: CIK Cell Transfusion Plus Gefitinib As Second Or Third-Line Treatment for Advanced Adenocarcinoma Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Kunming Medical University (Other)
Responsible Party: Principal Investigator, Song Xin, Chief of the Department of Cancer Biotherapy Center, The Third Affiliated Hospital of Kunming Medicine University, Kunming Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIK plus gefitinib
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; CIK; Gefitinib; Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Gefitinib combination with CIK cell immunotherapy
  Interventions: Drug: Group A:cytokine-induced killer cell +gefitinib
- Group B (Active Comparator): Gefitinib alone
  Interventions: Drug: Group B:Gefitinib

INTERVENTIONS:
Drug: Group A:cytokine-induced killer cell +gefitinib — CIK cells: intravenous infusions; D14-16; one cycle every month,at least 6 cycles;Gefitinib treated with 250mg for daily oral administration in the absence of disease progression or unacceptable toxicity.
  Arms: Group A
Drug: Group B:Gefitinib — Gefitinib treated with 250mg for daily oral administration in the absence of disease progression or unacceptable toxicity
  Arms: Group B

SUMMARY:
Lung cancer is the most common cancer worldwide, non-small cell lung cancer (NSCLC) comprises about 85% of all lung cancer cases, which is the leading cause of cancer mortality, and adenocarcinoma is the most prevalent subtype. Gefitinib showed lower efficiency of treatment as second or third-line in patients with advanced adenocarcinoma NSCLC. It is necessary to further improve the efficiency of treatment in patients with advanced NSCLC. Immunotherapy with cytokine-induced killer cells (CIK) may improve tumor control and survival, as well as a better quality of life. This study is to evaluate the efficacy of Autologous CIK Transfusion plus Gefitinib for advanced, recurrence, metastatic adenocarcinoma NSCLC.

DETAILED DESCRIPTION:
Lung cancer is the most common cancer worldwide, non-small cell lung cancer (NSCLC) comprises about 85% of all lung cancer cases, which is the leading cause of cancer mortality, and adenocarcinoma is the most prevalent subtype. The epidermal growth factor receptor (EGFR) adenosine triphosphate-competitive tyrosine kinase inhibitors gefitinib showed success in the treatment of advanced adenocarcinoma NSCLC following the failure of front-line chemotherapy. However, the efficiency of treatment as second or third-line in patients with advanced adenocarcinoma NSCLC is also low. It is necessary to further improve the efficiency of treatment in patients with advanced NSCLC. Biological treatment is an effective adjuvant treatment in comprehensive cancer treatment. Immunotherapy with cytokine-induced killer cells (CIK) characterized as fast amplification, strong anti-cancer activity and broad anti-tumor spectrum, this effect may improve tumor control and survival, as well as a better quality of life. This study is to evaluate the efficacy of Autologous CIK Transfusion plus Gefitinib for advanced, recurrence, metastatic adenocarcinoma NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 80 years
* Histologically or cytologically proven advanced adenocarcinoma non-small-cell lung cancer
* Life expectancy more than 12 weeks
* Not received EGFR agent or cell immunotherapy before entry into this study
* World Health Organization- Eastern Cooperative Oncology Group Performance Status 0-3
* Gefitinib as the second or third line therapy
* More than 4 weeks must have completion of the last dose of chemotherapy, radiation therapy, investigational therapy and patients must adequately recover from these effects
* Disease measurable
* Patients must have adequate organ and marrow functions as defined below: white blood cells: more than 3.0×109/L, Neutrophils: more than 1.5×109/L, Platelets: more than 75×109/L, Hemoglobin more than 80g/L, Serum total bilirubin less than 1.25 folds of the upper normal limit (ULN), Serum glutamic-oxal (o) acetic transaminase: less than 2.5×ULN, Serum glutamate pyruvate transaminase: less than 2.5×ULN, Serum creatinine: less than 1.25×ULN, Blood urea nitrogen: less than 2×ULN.
* Pregnancy test: the test of women of child-bearing period must be negative before entry into this study
* Subject must have good compliance and voluntarily to sign a written informed consent

Exclusion Criteria:

* Acute infection
* Uncontrolled concurrent illness: hypersensitiveness, asthma, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, serious heart valve disease
* Psychiatric illness, pharmacological dependence, or other situation that would limit compliance with study requirements
* History of other neoplasms
* Coagulation disorder and bleeding tendency
* Pertinacious hypertension（systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg) after aggressive therapy
* Brain metastasis with symptomatic
* Severe liver dysfunction
* Autoimmune disease (e.g. systemic lupus erythematosus, rheumatoid arthritis, thyroadenitis, et al )
* Patients who diagnosed as virus hepatitis, syphilis or HIV, or other infectious diseases
* Employment of corticosteroids or other immunodepressive hormone therapies
* With main organs transplantation
* Pregnant or lactating women
* Known or suspected in patients with severe hypersensitivity to CIK or gefitinib or to any other component of gefitinib
* Patients receiving any other investigational agents in 30 days or prepare to participate in other investigation in the clinical period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-11 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to 2 years

SECONDARY OUTCOMES:
Overall survival | up to 3 years

OTHER OUTCOMES:
Quality-of-life | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Xin Song, MD, Study Chair — The Third Affiliated Hospital of Kunming Medicine University
Locations (1):
- Department of Cancer Biotherapy Center, The Third Affiliated Hospital of Kunming Medicine University, Kunming, Yunnan, China